CLINICAL TRIAL: NCT06792604
Title: "Host Genome Methylation: a Screening Tool in Anal Cancer Detection"
Brief Title: Host Genome Methylation: a Screening Tool in Anal Cancer Detection
Acronym: AMethysT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP241033
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Anal Cancer
Keywords: HIV; MSM; Solid organ transplant; Vulvar lesions; Vulvar cancer
MeSH Terms: conditions — Anus Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Intervention Model Description: This study focuses on diagnostic and prognostic research for high-grade precancerous anal lesions. It is a prospective, single-centre, diagnostic and prognostic cohort study.
  Follow-up will vary depending on the HPV 16 result, but there is only one arm: cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort (Other): Patient HPV16 + at inclusion :
  * Cytological analysis of the smear
  * Referral to proctology (recommendation): Standard proctological examination Additional self-samples will be taken at 1 year (M12), 2 years (M24) and 3 years (M36 - end of follow-up) during a visit as part of standard care Questionnaire carried out at 1 year (M12), 2 years (M24) and 3 years (M36 - end of follow-up) during a visit as part of standard care
  And if cytology positive or if anal symptoms :
  * Standard proctological examination
  * Anal smear at clinician's discretion (virological analysis)
  * Anal biopsy if necessary (cytological analysis)
  * AHR (high-resolution anoscopy)
  Patient HPV16 - at inclusion :
  * Additional self-sampling at 3 years during a visit as part of standard care
  * Questionnaire carried out at 3 years during a visit as part of standard care And if anal symptom
  * Standard proctological examination, Anal smear, AHR at clinician's discretion
  * Anal biopsy if necessary
  Interventions: Device: Anal self-sampling (smear); Behavioral: HPV questionnaire

INTERVENTIONS:
Device: Anal self-sampling (smear) — Anal self-sampling (smear) at M12, M24 and M36 (each year) for HPV16+ patients at M0 and anal self-sampling (smear) at M36 for HPV16- at M0
Behavioral: HPV questionnaire — HPV questionnaire at each visit M0, M12, M24 and M36 for HPV16-positive patients at M0 and HPV questionnaire at each visit M0, 4 and M36 for HPV16-negative patients

SUMMARY:
In January 2023, the first recommendations for anal cancer screening were issued by the French National Society of Coloproctology (SNFCP). These were the world's first national recommendations for anal cancer screening for at-risk patients, not limited to people living with HIV. They are based on screening for papillomavirus type 16 (HPV16) as the first line of defence, followed by reflex cytology in the event of a positive HPV16 smear and a proctological examination. In the event of abnormal cytology or proctological examination, high-resolution anoscopy (HRA) should be performed, but access to it is limited by the number of proctologists with the expertise to carry out this examination and the cost of the equipment. The development of biological markers could enable only patients at high risk of high-grade dysplasia/anal cancer to be referred for HRA.

As part of the AIN3 cohort, we demonstrated that the markers ZNF582 and ASCL1, studied on anal smears taken when patients were included in the cohort, showed a significantly higher level of methylation in patients who subsequently progressed to anal cancer.

The aim of this project is to test, in real-life conditions, the contribution of these methylation markers in the triage of asymptomatic patients eligible for anal cancer screening according to the SNFCP guidelines (MSM over 30 years of age living with HIV, women with a history of vulvar lesions or vulvar, women patients who have had a solid organ transplant for more than 10 years and extension to men patients who have had a solid organ transplant for more than 10 years).

DETAILED DESCRIPTION:
I. Current state of knowledge on the pathology

In 2020, 30,000 cases of squamous cell carcinoma of the anus were reported worldwide. These cancers affect women in 2/3 of cases. They are fairly rare in the general population, with an age-standardised incidence rate of 0.35 per 100,000 person-years (p.a.) in men and 0.57 in women.

The population of men who have sex with men (MSM) living with HIV is at greater risk of anal cancer: studies in 2012 reported an 80-fold increase in the relative risk compared with the non-HIV-infected male population. This population is also more exposed to anal HPV infections, which adds to the dysimmunity associated with HIV infection. As a result, this population was already the subject of specific recommendations concerning anal canal cancer screening based on cytology. A recent meta-analysis has stratified the risk of anal cancer in different populations. It confirms the excess risk of anal cancer in the MSM population living with HIV (up to 100 per 100,000 pa in MSM living with HIV aged over 45).

It has also identified other groups at risk of anal cancer. A higher incidence rate of anal cancer in women who have already had cervical or vulvovaginal cancer is clearly established. But this meta-analysis by Clifford et al. shows a different stratification of anal cancer risk according to the type of previous HPV-induced cancer. Thus, the incidence rate of anal cancer is highest in the case of a history of vulvar cancer, equal to 50 per 100,000 pa, whereas it is close to 10 per 100,000 pa in the case of a history of vaginal or cervical cancers. Another group at risk of anal cancer is made up of immunosuppressed people not infected with HIV, and in particular solid transplant recipients, with different incidence rates of anal cancer depending on the type of transplant and above all the time since the transplant.

Overall, incidence rates of anal cancer, regardless of sex, are higher in high-income countries. In 2018, 1,532 new cases of anal cancer were reported in women in France, corresponding to an incidence rate of 2.4 per 100,000 woman-years, and 479 new cases in men, corresponding to an incidence rate of 0.8 per 100,000 man-years. As in many high-income countries, an overall increase in the incidence of this cancer has been observed in France, both in women (+3.4% and +5.7% between 1990 and 2018 and between 2010 and 2018 respectively) and in men (+1.5% and +3.3% between 1990 and 2018 and between 2010 and 2018 respectively). Trends by age for anal cancer show an increase in the number of cases, mainly in women aged 50 and 60.

Analysis of human genome methylation in anal swabs is a promising biomarker for anal cancer risk. Methylation is an epigenetic physiological phenomenon that regulates the expression of certain genes. The viral oncoproteins E6 and E7 of high-risk oncogenic HPVs (notably HPV16) have been shown to induce activation or increased expression of the cellular enzymes responsible for these methylation phenomena. As a general rule, hypermethylation of gene promoters leads to their inactivation. Repression of genes involved in the antiviral or anti-tumour response may contribute to immune escape, whereas hypermethylation inducing repression of tumour suppressor genes favours the cancerous process.

With regard to anal cancer, two studies demonstrated that the methylation markers previously developed for the cervix were not discriminatory for anal cancer. Subsequently, cross-sectional analysis of anal biopsies at different stages (normal cytology, low-grade or high-grade lesions, cancer) has revealed methylation markers specific to anal carcinogenesis in anal biopsies (invasive tissue sampling).

These markers are extremely promising, and methylation could therefore constitute a robust predictive marker of progression to an invasive lesion, and would therefore be a decisive factor in the decision of invasive treatment versus surveillance.

II. State of knowledge on reference procedures

The evolution of anal pre-cancerous lesions is less well described than that of cervical lesions due to the absence of screening programmes to date.

For the first time, the American ANCHOR study of nearly 5,000 PLHIV demonstrated the impact of treatment of high-grade lesions, with a 57% reduction in the rate of cancer in the treated arm (incidence 173 per 100,000 pa vs 402 per 100,000 pa in the simple surveillance arm). Following this study, recommendations for screening for precancerous anal lesions in asymptomatic at-risk populations are beginning to emerge.

In January 2023, the French National Society of Colo-Proctology (SNFCP) issued recommendations for anal cancer screening of asymptomatic individuals in three at-risk populations: MSM living with HIV aged over 30, women with a history of pre-cancerous lesion or cancer of the vulva and women who have received a solid organ transplant for more than 10 years. These recommendations target populations with an incidence of anal cancer greater than 40 per 100,000 pa according to the meta-analysis by Clifford et al. In this context, screening for anal cancer is based on primary HPV16 screening, in particular by anal self-sampling and, if positive, an anal smear for cytology and a standard proctology examination. In the event of abnormal cytology, patients will be referred for a proctology consultation with high-resolution anoscopy (HRA).

There are few proctologists in France who carry out AHR examinations, and waiting times for consultations are already very high. The major stumbling block to the introduction of anal cancer screening is the anticipated worsening of the overcrowding of AHR examinations and proctology consultations. For example, a recent meta-analysis reported a prevalence of 27% to 35% of HPV16 infection in the anal region of MSM living with HIV. The development of triage tools enabling only those patients most at risk of high-grade anal dysplasia to be referred for this examination is therefore crucial.

The aim of this new study is to validate the predictive capacity of anal smear methylation markers for screening patients at risk of progressing to high-grade dysplasia and to define appropriate thresholds in this sample, including patients targeted by the new SNFCP screening recommendations and therefore with no history of AIN3 lesions.

III. Hypothesis

This study is based on the hypothesis that the level of methylation of the markers ASCL1 and ZNF582 will be predictive of the risk of asymptomatic patients developing high-grade anal lesions and therefore anal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age ≥ 18 years)
2. Eligible for anal cancer screening according to the SNFCP guidelines (with extension to men who have received solid organ transplants for more than 10 years):

   * MSM (men who have sex with men) aged over 30 living with HIV
   * Patients who have received a solid organ transplant for more than 10 years
   * Women with a history of vulvar lesions or vulvar cancer

Non-inclusion Criteria:

1. Proctological follow-up for a current high-grade anal lesion or cancer
2. Pregnant or breastfeeding women
3. Subject deprived of liberty or under legal protection
4. Non-affiliation with social security system
5. Refusal to participate expressed by the patient

Exclusion Criteria :

1) Refusal of anal self-sampling on inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — MSM (men who have sex with men) over 30 years old living with HIV Women with a history of vulvar lesions or vulvar cancer
Enrollment: 770 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2028-11-22 (Estimated); Study Completion 2028-11-22 (Estimated)

PRIMARY OUTCOMES:
High- grade anal lesion at 3 years | 3 years after Inclusion
  Analyse if methylation markers on an initial anal self sample (M0) could predict high grade anal lesion at M3

SECONDARY OUTCOMES:
HSIL cytology on the anal self-sample at 3 year in HPV 16 negative patients at M0 | 3 years after Inclusion
  Evaluation of the predictive characteristics of methylation markers on a first anal self-sampling for the absence at 3 years of high grade anal lesions (HSIL) in patients considered at risk of anal cancer according to the SNFCP recommendations after a first self-sampling in HPV 16 negative patients at M0.
High grade anal lesion in HPV 16 positive patients at M0 | 1 year, 2 years, 3 years after inclusion
  Evaluation of the time dependant predictive characteristics of methylation markers to predict the evolution of HPV 16+ patients at M0 towards high grade anal lesions (HSIL) in patients considered to be at risk of anal cancer according to the SNFCP recommendations.
Diagnostic properties of methylation in HPV 16-positive patients at M0 | M0
  Validation of methylation as a diagnostic tool for high-grade lesions in HPV 16+ patients
Persistance of HPV infection | 4 years after the inclusion of the first patient
  Time to HPV negativation
Time for HPV16 clearance | 3 years after Inclusion
  Time from initial anal self sample HPV16 + to first sample HPV16- :
  Analyse factors associated with time for HPV 16 clearance.
Incidence of high grade Anal lesions | 3 years after Inclusion
  Prevalence and incidence of pre-cancerous and cancerous anal lesions
Number of protocol-eligible patients refusing to participate | 4 years after the inclusion of the first patient
  Acceptability and applicability of the different stages of the anal cancer screening programme in a tertiary centre with expertise in the subject
Methylation levels | 1 year, 2 years, 3 years after inclusion
  Evolution of methylation over time
Rate of patients with a follow-up in accordance with French national recommendations after HPV16 positive self anal sampling | 4 years after the inclusion of the first patient
  Acceptability and applicability of the different stages of the anal cancer screening programme in a tertiary centre with expertise in the subject

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Cardiovascular Surgery and Transplantation Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Dermatology Department, Paris, Île-de-France Region
  - Gynecology and Obstetrics Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Hepato-Gastroenterology, Digestive Oncology, and Proctology Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Infectious and Tropical Diseases Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Nephrology Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Pathological Anatomy and Cytology Department Bichat-Claude Hospital, Paris, Île-de-France Region
  - Pulmonology B and Lung Transplantation Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region
  - Virology Department Bichat-Claude Bernard Hospital, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided